CLINICAL TRIAL: NCT02996513
Title: Assessing Model Parameters for Applying the Retinol Isotope Dilution (RID) Method in Preschool Nigerian Children Living in an Area With a High Malaria Burden
Brief Title: Assessing Model Parameters for Applying the Retinol Isotope Dilution (RID) Method
Acronym: SUPERKID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: University of Ibadan (Other); Newcastle University (Other); University of California, Davis (Other); Penn State University (Other); HarvestPlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WageningenU
Record Dates: First submitted 2016-11-11; First posted 2016-12-19 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Vitamin A Deficiency; Malaria; Inflammation
Keywords: Vitamin A status; Retinol Isotope Dilution; Nigeria; Preschool children; Malaria; Inflammation
MeSH Terms: conditions — Vitamin A Deficiency; Malaria; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Retinol Isotope dilution (RID) (Experimental): A once-off dose of 0.4 mg 13C4-retinyl acetate will be administered to subjects as a capsule
  Interventions: Other: Retinol Isotope Dilution (RID)

INTERVENTIONS:
Other: Retinol Isotope Dilution (RID) — 13C-retinyl acetate will be administered to subjects in order to assess their body retinol pools

SUMMARY:
For assessing body retinol pools in preschool children, it is recommended that a blood sample is taken 14-21 days after isotope dosing. During this period, dietary intake of vitamin A should be controlled. Shortening of this period as has been validated for adults would reduce the burden for the children as well as improve research efficiency. The aim is to validate a 4-day protocol for assessing body retinol pools in preschool children by modelling data derived by retinol isotope dilution (RID) method. Venous blood samples will be collected of 60 children 4 days after dosing of 0.4 mg 13C-labeled retinyl acetate. A second venous blood sample will be collected at 6, 8, 12 hrs; and 1, 2, 4, 7, 11, 16, 22 and 28 days after dosing in subgroups of 6 children, randomly divided over the 10 additional time points. Body retinol pools will be modelled, and the time point at which a parsimonious model applies (presumably at day 4) will be assessed.

DETAILED DESCRIPTION:
For assessing body retinol pools in preschool children, it is recommended that a blood sample is taken 14-21 days after isotope dosing. During this period, dietary intake of vitamin A should be controlled. Shortening of this period as has been validated for adults would reduce the burden for the children as well as improve research efficiency. The aim is to validate a 4-day protocol for assessing body retinol pools in preschool children by modelling data derived by retinol isotope dilution (RID) method. A secondary aim is to compare body retinol pools between children with and without inflammation and to assess the effect of asymptomatic malaria on model parameters. Preschool children (n=60), 36-59 months of age, residing in Telemu, Osun State, Nigeria will be recruited for the study. The study design is an observational pre/post study, for which body retinol pools will be measured using the RID method. Venous blood samples will be collected of all children 4 days after dosing of 0.4 mg 13C-labeled retinyl acetate. A second venous blood sample will be collected at 6, 8, 12 hrs; and 1, 2, 4, 7, 11, 16, 22 and 28 days after dosing in subgroups of 6 children, randomly divided over the 10 additional time points. Children presenting with asymptomatic malaria will be treated, and a convenience subsample (n=10) will undergo a second assessment of body retinol pools determined with a venous blood collection on day 4 post-dosing only. Body retinol pools will be modelled, and the time point at which a parsimonious model applies (presumably at day 4) will be assessed. Presence of asymptomatic malaria and markers of inflammation will be assessed in all children at all time points. Body retinol pools and model parameters between subgroups of children with and without asymptomatic malaria and/or inflammation will be compared. Pre/post comparisons of body retinol pool estimates will be done for the follow up subsample.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy
* Between 36 and 59 months of age
* Living in the community of Telemu, Osun State, Nigeria, or its neighbouring communities

Exclusion Criteria:

* Active or recent disease with a potential effect on study outcome
* Hb concentration <70 g/dL
* Mental state that is incompatible with participation in the study
* Recent exposure to 13C-retinol stable isotopes
* Unwillingness to participate by verbal or physical expression

Ages: 36 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Vitamin A status | 28 days
  Body retinol pool

SECONDARY OUTCOMES:
Prevalence of malaria (plasmodium falciparum) | 28 days
  Percentage of children with malaria (Plasmodium falciparum) as determined by a rapid test (CareStart Malaria HRP2) and confirmed by PCR.
Prevalence of inflammation | 28 days
  Percentage of children with C-reactive protein (CRP) >5 mg/L and/or alpha-glycoprotein (AGP) >1 g/L
Serum retinol | 28 days
  Serum concentration of retinol (HPLC)
Blood haemoglobin concentration | 28 days
  Haemoglobin concentration (Quikread)
Ferritin concentration | 28 days
  Serum concentration of ferritin (ELISA)
Soluble transferrin receptor concentration | 28 days
  Serum concentration of soluble transferrin receptor concentration (ELISA)
Retinol binding protein | 28 days
  Serum concentration of retinol binding protein (ELISA)

OTHER OUTCOMES:
Body weight | Baseline
  Body weight will be measured to the nearest 0.1 kg with a weighing scale
Dietary intake of energy, protein, fat, carbohydrates, vitamins and minerals | Baseline
  Group mean intake of macronutrients and micronutrients, assessed by 24h recall
Body length | Baseline
  Body length will be measured to the nearest 1 cm with a stadiometer

CONTACTS AND LOCATIONS:
Overall Officials: Alida Melse-Boonstra, PhD, Principal Investigator — Wageningen University
Locations (1):
- University of Ibadan, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: No